CLINICAL TRIAL: NCT04588194
Title: Romiplostim in Combination With Low-dose Rituximab and High-dose Dexamethasone as Frontline Treatment for Immune Thrombocytopenia
Brief Title: Romiplostim, Rituximab and Dexamethasone as Frontline Treatment for Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Gomez Almaguer (Other)
Responsible Party: Sponsor-Investigator, David Gomez Almaguer, David Gómez Almaguer, Hospital Universitario Dr. Jose E. Gonzalez
Organization: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hospital Universitario
Record Dates: First submitted 2020-01-30; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Immune Thrombocytopenia; Thrombotic Thrombocytopenic Purpura
Keywords: thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombotic Thrombocytopenic; Thrombocytopenia | interventions — romiplostim; Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Romiplostim, Rituximab, Dexamethasone (Experimental): Each patient will receive Rituximab 100 mg weekly days 1, 7, 14, 21, Romiplostim 2mcg/Kg subcutaneously weekly days 1, 7, 14, 21 and Dexamethasone 40 mg IV/PO days 1-4.
  Interventions: Drug: Romiplostim; Drug: Rituximab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Romiplostim — Romiplostim 2mcg/Kg subcutaneously weekly days 1, 7, 14, 21
Drug: Rituximab — Rituximab 100 mg weekly days 1, 7, 14, 21
Drug: Dexamethasone — 40 mg IV/PO days 1-4

SUMMARY:
The purpose of this study is to determine the response rate and response duration with the combination of low-dose rituximab, romiplostim and high-dose dexamethasone.

DETAILED DESCRIPTION:
Immune thrombocytopenia is an autoimmune disorder characterized by formation of autoantibodies against platelet antigens leading platelet destruction.

Corticosteroids increase the platelet count in about 80 percent of patients. However, many patients have a relapse when the dose of corticosteroid is reduced. Debilitating side effects are common in patients who require long-term corticosteroid therapy to maintain the platelet count. Romiplostim, it is a small molecule agonist of the c-mpl (TpoR) receptor, which is the physiological target of the hormone thrombopoietin, has been shown to be effectively raise the platelet count in adult patients (aged 18 years and over) who have had their spleen removed or where splenectomy is not an option and have received prior treatment with corticosteroids or immunoglobulins, and these medicines did not work (refractory ITP). There are a few case reports where romiplostim an option as first line treatment for IT.

The purpose of this study is to determine the response rate and response duration with the combination of rituximab (100 mg weekly four weeks), romiplostim (2mcg/Kg four weekly) and high-dose dexamethasone (40mg PO days 1-4) in untreated adult patients with <30*109/L platelet count diagnosed with immune thrombocytopenia.

A complete response is defined as an increase in platelet counts to >150×109/L on two consecutive occasions. A clinical response is defined as an increase in the platelet count between >30×109/L on two consecutive measures and no bleeding. Duration of response is considered from the day of the initial administration to the first time of relapse (platelet count <30×109/L) or to time of analysis Patients will be evaluated each week during 4 weeks and then every month for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed immune thrombocytopenia (IT) Platelet count less than 30,000/mm3 on two occasions.
* Subject ≥ 16 years
* Subject has signed and dated written informed consent.

Exclusion Criteria:

* Previous treatment (only corticosteroids at dose or prednisone equivalent of 300 mg)
* Performance status above or equal to 2.
* Pregnancy and lactation
* Previous splenectomy
* Connective tissue disease
* Autoimmune hemolytic anemia
* Relapse
* Active infection, sepsis or fever
* Positive for hepatitis B virus or hepatitis C virus or human immunodeficiency virus.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 28 days
  Platelet counts to >30×109/L on two consecutive occasions

SECONDARY OUTCOMES:
Complete Response | 28 days
  Platelet counts to >100×109/L on two consecutive occasions

CONTACTS AND LOCATIONS:
Overall Officials: David Gómez, MD, Principal Investigator — Hospital Universitario J. Eleuterio González
Locations (1):
- Servicio de Hematología, Hospital Universitario "Dr. José Eleuterio González", Universidad Autónoma de Nuevo León, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomez-Almaguer D, Herrera-Rojas MA, Jaime-Perez JC, Gomez-De Leon A, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Tarin-Arzaga L, Hernandez-Reyes J, Ruiz-Arguelles GJ. Eltrombopag and high-dose dexamethasone as frontline treatment of newly diagnosed immune thrombocytopenia in adults. Blood. 2014 Jun 19;123(25):3906-8. doi: 10.1182/blood-2014-01-549360. Epub 2014 May 6. PMID 24802773
- [Result] Gomez-Almaguer D, Tarin-Arzaga L, Moreno-Jaime B, Jaime-Perez JC, Ceballos-Lopez AA, Ruiz-Arguelles GJ, Ruiz-Delgado GJ, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Sanchez-Cardenas M. High response rate to low-dose rituximab plus high-dose dexamethasone as frontline therapy in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2013 Jun;90(6):494-500. doi: 10.1111/ejh.12102. Epub 2013 Apr 2. PMID 23470153
- [Result] Cooper N, Terrinoni I, Newland A. The efficacy and safety of romiplostim in adult patients with chronic immune thrombocytopenia. Ther Adv Hematol. 2012 Oct;3(5):291-8. doi: 10.1177/2040620712453596. PMID 23616916
- [Result] Vishnu P, Aboulafia DM. Long-term safety and efficacy of romiplostim for treatment of immune thrombocytopenia. J Blood Med. 2016 May 25;7:99-106. doi: 10.2147/JBM.S80646. eCollection 2016. PMID 27307776